CLINICAL TRIAL: NCT01620593
Title: Phase II, Randomized, Placebo Controlled, Double Blind, Prospective Study of Castration Compared to Castration Plus Metformin as First Line Treatment for Patients With Advanced Prostate Cancer.
Brief Title: Castration Compared to Castration Plus Metformin as First Line Treatment for Patients With Advanced Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CTRC 10-21; HSC20110273H (Other: UTHSCSA IRB)
Record Dates: First submitted 2012-05-31; First posted 2012-06-15 (Estimated); Results first posted 2018-05-22 (Actual); Last update posted 2018-05-23 (Actual); Status verified 2016-09

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Metformin; Castration therapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Metabolic consequences including development of hyperinsulinemia and insulin resistance using metformin compared to placebo in men on castration therapy.
  Interventions: Drug: Placebo
- Metformin (Active Comparator): Metabolic consequences including development of hyperinsulinemia and insulin resistance using metformin compared to placebo in men on castration therapy. In the rare case where a patient may not tolerate 500 mg three times a day, he may remain on the study taking only 500 mg twice a day.
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Placebo — All eligible subjects will be randomized in a 1:l manner to receive a bottle containing sufficient 500mg tablets of placebo after castration, blinded to the patient and the study team.
  Arms: Placebo
Drug: Metformin — All eligible subjects will be randomized in a 1:l manner to receive a bottle containing sufficient 500mg tablets of metformin after castration, blinded to the patient and the study team.
  Arms: Metformin

SUMMARY:
Prostate cancer is the most common non-cutaneous cancer in men. Patients with recurrent or metastatic prostate cancer are treated with androgen-deprivation therapy, often termed castration therapy. While the short and medium term benefits of castration are clear in relation to therapeutic efficacy in patients with prostate cancer, it is now appreciated that the resulting hypogonadism associated with castration is responsible for adverse consequences or metabolic syndrome that include increase in body mass index (BMI) and fat mass, hyperinsulinemia and insulin resistance, hyperlipidemia, reduced lean body mass (LBM) and muscle strength, osteoporosis, sexual dysfunction, poor quality of life and higher cardiovascular mortality. Lower testosterone levels in men independently predict the development of metabolic syndrome. Low testosterone levels in men are associated with insulin resistance and diabetes. Metformin is commonly prescribed for the treatment of type II diabetes because it lowers both glucose and insulin levels. Studies show preliminary evidence that metformin might have both antineoplastic and chemopreventative activity. Castration therapy decreases insulin sensitivity, adversely alters lipid profiles and results in weight gain, and it may be associated with a greater incidence of diabetes and cardiovascular disease. Little is known about the optimal strategy to mitigate the adverse metabolic effects of castration in men with prostate cancer. The rationale for using metformin in castrated men with advanced prostate cancer stems from the observation that castration therapy is associated with the metabolic syndrome, hyperinsulinemia and insulin resistance. Furthermore, reports that hyperinsulinemia stimulates insulin receptor expression on prostate cancer leading to tumor growth and development of castrate resistant prostate cancer suggest metformin through its activation of the AMPK-LKBI pathway reduces liver gluconeogenesis secondarily decreasing insulin levels may circumvent tumor growth and resistance to castration therapy. More importantly, evidence that metformin inhibits the mTOR pathway implicates an added therapeutic benefit as an anti-cancer agent.

ELIGIBILITY:
Inclusion Criteria:

(Eligible subjects must meet one of the inclusion criteria 1-3 and all of items 4-6)

1. Men with metastatic prostate cancer that require castration therapy with either using an LHRH analogue or surgical castration are eligible. Complete androgen blockade using anti-androgen therapy prior to castration or up to 4 weeks following castration therapy is permitted to prevent disease flare. Thereafter anti-androgen therapy may continue or be discontinued based on treating physicians preference.

   OR
2. Any men with prostate cancer who are candidates for castration therapy despite no evidence of definite metastatic disease including patient with biochemical failure or 'rising PSA' are also permitted to enter study provided castration therapy is planned for a minimum of a year. Patients with biochemical failure prior to enrolment should have also have already received appropriate salvage therapy. Men with prostate cancer who have already started castration therapy are also permitted to enter study provided castration therapy was initiated within one month of study entry.

   OR
3. Men with prostate cancer previously treated with castration therapy for management of localized prostate cancer in the adjuvant setting or in combination with radiation therapy are permitted to enter study provided they currently have known metastatic disease and have non-castrate testosterone levels (Testosterone > 50 ng/dL).
4. An ECOG performance status of 0-2.
5. Patients will need to have documentation of metastatic disease in bone and/or soft tissue, and a baseline PSA of ≥ 5 ng/ml. If patients have already had castration therapy, their baseline PSA value will be reflective of the value prior to castration. Patients with biochemical failures, with rising PSA (baseline PSA does not need to be ≥ 5 nglml to be eligible), without metastatic disease are also eligible if castration therapy is indicated for minimum of 7 months and for these patients any PSA value is permitted.
6. Patients must have provided informed consent, be willing to have blood specimens taken, and exhibit no severe other medical or psychiatric problems.

Exclusion Criteria:

1. Patients with severe medical or psychiatric diseases are INELIGIBLE. (Patients with stable chronic diseases such as high cholesterol or hypertension ARE eligible.) Examples of problems that would make patients INELIGIBLE include severe heart failure, or hypoxia due to severe lung disease.
2. Patients with clinical or biochemical evidence of renal failure or liver failure are INELIGIBLE. Creatinine and bilirubin needs to be less than or equal to 1.3~up per limit of normal (ULN), and ASTIALT less than or equal to 2.5 x ULN unless liver metastasis is present then up to 5 X ULN permitted).
3. Patients already receiving metformin or anti-diabetic medications are INELIGIBLE.
4. If any patient develops symptomatic diabetes requiring drug therapy, he must receive such a therapy, which may include metformin. This must be documented, and the patient will not continue on the study.
5. Patients with important infections requiring antibiotics are INELIGIBLE, but patients who acquire minor infections while on the study may remain on the study.
6. Alcohol abuse problems make patients INELIGIBLE. Patients need to be consuming less than or equal to 14 units of alcohol weekly.
7. Patients with history or evidence of lactic acidosis or metabolic acidosis will be excluded.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2011-04; Primary Completion 2016-07 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Devalingam Mahalingam, MD, PhD, Principal Investigator — University of Texas Health Science Center San Antonio
Locations (1):
- Cancer Therapy and Research Center University of Texas Health Science Center San Antonio, San Antonio, Texas, United States

REFERENCES:
- [Derived] Roy S, Malone S, Grimes S, Morgan SC. Impact of Concomitant Medications on Biochemical Outcome in Localised Prostate Cancer Treated with Radiotherapy and Androgen Deprivation Therapy. Clin Oncol (R Coll Radiol). 2021 Mar;33(3):181-190. doi: 10.1016/j.clon.2020.09.005. Epub 2020 Sep 29. PMID 32994091
- See also: Abstract in Journal of Clinical Oncology — http://ascopubs.org/doi/abs/10.1200/JCO.2017.35.15_suppl.e16502

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo and Castration: Metabolic consequences including development of hyperinsulinemia and insulin resistance using metformin compared to placebo in men on castration therapy.
  Placebo and Castration: All eligible subjects will be randomized in a 1:l manner to receive a bottle containing sufficient 500mg tablets of metformin or placebo, blinded to the patient and the study team.
- Metformin and Castration: Metabolic consequences including development of hyperinsulinemia and insulin resistance using metformin compared to placebo in men on castration therapy. In the rare case where a patient may not tolerate 500 mg three times a day, he may remain on the study taking only 500 mg twice a day.
  Metformin and Castration: All eligible subjects will be randomized in a 1:l manner to receive a bottle containing sufficient500mg tablets of metformin or placebo, blinded to the patient and the study team.
Period: Overall Study
Arm/Group | Placebo and Castration | Metformin and Castration
Started | 21 | 20
Completed | 17 | 19
Not Completed | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo and Castration | Metformin and Castration | Total
Number analyzed (Participants) | 17 | 19 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 19 | 36
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 17 | 19 | 36
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17 | 19 | 36

OUTCOME MEASURES:

1. Primary Outcome: Metabolic Syndrome
Description: Compare both cohorts of castrated men (metformin vs. placebo) with regard to metabolic consequences of castration therapy:change in weight.
Time Frame: Change from 0 weeks to 28 weeks
Population: Only subjects that completed the study were analyzed
Measure: Mean (Full Range); unit: kilograms
Arm/Group | Placebo and Castration | Metformin and Castration
Number analyzed (Participants) | 17 | 19
kilograms | 0 [0 to 0] | 0 [0 to 0]

2. Primary Outcome: Metabolic Syndrome Waist Circumference
Description: Compare both cohorts of castrated men (metformin vs. placebo) with regard to metabolic consequences of castration therapy:change in waist circumference.
Time Frame: Change from 12 to 28 weeks
Measure: Mean (Full Range); unit: centimeters
Arm/Group | Placebo and Castration | Metformin and Castration
Number analyzed (Participants) | 17 | 19
centimeters | 40.52 [29.5 to 47.5] | 41.14 [30.25 to 50.0]
Statistical Analysis 1: Comparison: Placebo and Castration vs Metformin and Castration; Test type: Superiority — t-test; p < 0.05, t-test, 2 sided

3. Secondary Outcome: PSA Response
Description: Complete Response for PSA measure was defined as a PSA less than or equal to 4 ng/ml or undetectable value at 7 months.
Time Frame: 28 weeks
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Placebo and Castration | Metformin and Castration
Number analyzed (Participants) | 17 | 19
ng/ml | 58.2 (193.43) | 8.36 (18.35)

4. Secondary Outcome: Treatment Failure
Description: Progression time from randomization to the earliest disease progression defined as an increase of 20% or more as per RECIST criteria. Patients will not be removed from protocol treatment for PSA progression alone in the first 12 weeks on this study. Further rise in PSA even in the absence of deterioration of pre-existing lesions will constitute treatment failure. Adverse event leading to withdrawal related to metformin or placebo or castration treatment. Death from any cause. Patients unwillingness to continue. Patient's non-compliance with taking the study intervention - 50% or higher.
Time Frame: 1 year
Population: Outcome was not measured
Arm/Group | Placebo and Castration | Metformin and Castration
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Number of Participants With Adverse Events
Description: The safety and tolerability of metformin with castration therapy as compared to castration therapy alone as measured by the number of subjects experiencing adverse events using CTCAE (common terminology criteria for adverse events) version 4 criteria. Grades are assigned to each adverse event where:
  Grade 1 is mild symptoms Grade 2 is moderate symptoms Grade 3 is severe or medically significant but not immediately life-threatening symptoms Grade 4 is life-threatening consequences, where urgent intervention is indicated Grade 5 is death related to the adverse event
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo and Castration | Metformin and Castration
Number analyzed (Participants) | 17 | 19
Participants
  Greater than or equal to 1 adverse event | 0 | 2
  Adverse event leading to treatment dose reduction | 0 | 7

ADVERSE EVENTS:
Arm/Group | Placebo and Castration | Metformin and Castration
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/19
Other Adverse Events (participants affected / at risk) | 2/17 | 8/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo and Castration (N=17) | Metformin and Castration (N=19)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 3 (3)
Muscle Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (3)
Increased Creatinine (Renal and urinary disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes